CLINICAL TRIAL: NCT04286282
Title: Neuroinflammation and Modulating Factors in Depression and HIV: The Growth Study-Group Therapy in HIV for Depression IN Uganda
Brief Title: Neuroinflammation and Modulating Factors in Depression and HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006374; K23MH121220 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Depression; HIV
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Active Comparator): The first 100 participants with HIV and depression will receive standard of care including SSRI therapy.
  Interventions: Other: Depression Standard of Care; Other: HIV Standard of Care
- Standard of Care + Group Support Psychotherapy (Experimental): The second 100 participants with HIV and depression will receive standard of care, including SSRI therapy, and group support psychotherapy.
  Interventions: Behavioral: Group Pyschotherapy; Other: Depression Standard of Care; Other: HIV Standard of Care
- Standard of Care (Non-Depressed) (Active Comparator): 100 participants with HIV and without depression will receive standard of care therapy for HIV and no depression treatment.
  Interventions: Other: HIV Standard of Care

INTERVENTIONS:
Behavioral: Group Pyschotherapy — Group psychotherapy
  Arms: Standard of Care + Group Support Psychotherapy
Other: Depression Standard of Care — Standard clinical care for depression, which may include the use of selective serotonin re-uptake inhibitors (SSRIs).
  Arms: Standard of Care; Standard of Care + Group Support Psychotherapy
Other: HIV Standard of Care — Standard clinical care for HIV

SUMMARY:
Determine if depression, which persists after depression treatment at 26 weeks, is associated with increased innate inflammation in a prospective cohort of HIV-infected Ugandans receiving SSRIs in which group psychotherapy is initiated.

DETAILED DESCRIPTION:
Depression in HIV is a complex co-morbidity with both social factors such as stigma as well as biologic components. Disruptions in neurotransmitters such as serotonin and catecholamines are known to cause depression. Inflammation caused by diseases such as stroke, diabetes, and HIV is associated with higher rates of depression. HIV causes inflammation throughout the body, but since the virus can cross the blood-brain-barrier, HIV can replicate in and target the brain causing neuroinflammation which predisposes depression. However the pathophysiology of the role of inflammation in comorbid depression and HIV is poorly understood.

1. Among depressed HIV-infected Ugandans, determine if the resolution of depression at 26 weeks of HIV therapy is improved with group psychotherapy.
2. In the same population determine if persistent depression is associated with higher levels of innate inflammation. Also, compare baseline and follow up inflammation among depressed compared to non-depressed control group.
3. Evaluate if viral suppression levels at 26 weeks are improved by group psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

For the depressed patient arm,

* Newly-presenting clinic patients (<3 months)
* Mild to Moderately-Severe Depressive Symptoms with PHQ-9 score >5 but <20
* Not suicidal (PHQ-9 question 9 score >2)
* Not receiving antiretroviral therapy (ART) at screening
* Outpatient, not requiring hospitalization

For the non-depressed patient arm,

* Newly-presenting clinic patients (<3 months)
* Not suicidal (PHQ-9 question 9 score >2)
* Not receiving antiretroviral therapy (ART) at screening
* Outpatient, not requiring hospitalization

Exclusion Criteria:

- No additional exclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lofgren, MD, Principal Investigator — University of Minnesota
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Standard of Care + Group Support Psychotherapy
Started | 62 | 47
Completed | 61 | 42
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Standard of Care + Group Support Psychotherapy | Total
Number analyzed (Participants) | 62 | 47 | 109
Age, Continuous [Mean (Full Range); unit: YEARS] | 29 [26 to 40] | 29 [25 to 37] | 29 [25 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 31 | 74
  Male | 19 | 16 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 62 | 47 | 109
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Health Questionnaire (PHQ)-9
Description: The Patient Health Questionnaire (PHQ)-9 is a 9-item survey measuring degree of depression severity over the previous 2 weeks. Items assess how often the patient has been bothered by specific symptoms and are rated on a scale of 0 (not at all) to 3 (nearly every day). Total score is an unweighted sum of the 9 item scores, with higher scores indicating greater depression severity.
  a score of 0-27 is possible. We aren't reporting subscales. A score of 5+ will screen positive for mild depression, and a score of 10+ is considered a positive to screen for moderate-severe depression.
  change between baseline and 3 months
Time Frame: 3 months
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Standard of Care + Group Support Psychotherapy
Number analyzed (Participants) | 62 | 47
units on a scale | 5 [2 to 7] | 7 [5 to 11]

2. Primary Outcome: Change in Patient Health Questionnaire (PHQ)-9
Description: The Patient Health Questionnaire (PHQ)-9 is a 9-item survey measuring degree of depression severity over the previous 2 weeks. Items assess how often the patient has been bothered by specific symptoms and are rated on a scale of 0 (not at all) to 3 (nearly every day). Total score is an unweighted sum of the 9 item scores, with higher scores indicating greater depression severity.
  a score of 0-27 is possible. We aren't reporting subscales. A score of 5+ will screen positive for mild depression, and a score of 10+ is considered a positive to screen for moderate-severe depression.
  change between baseline and 6 months
Time Frame: 6 months
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care | Standard of Care + Group Support Psychotherapy
Number analyzed (Participants) | 62 | 47
units on a scale | 7 [5 to 8] | 8 [6 to 11]

ADVERSE EVENTS:
Time Frame: Not collected
Description: Adverse events were not collected
Arm/Group | Standard of Care | Standard of Care + Group Support Psychotherapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT04286282/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT04286282/ICF_001.pdf